CLINICAL TRIAL: NCT03096626
Title: Association Between Depression and Iron Metabolism in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Yoshihiro Tsuji (Other)
Responsible Party: Sponsor-Investigator, Yoshihiro Tsuji, University of Hyogo, University of Hyogo
Organization: University of Hyogo (Other)
Other Study IDs: Uhyogo2
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Hemodialysis
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study assesses the association of depression symptoms and iron metabolism in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
The Beck Depression Inventory (BDI), second version, was used to quantify the levels of depression. Mean age, duration of HD, hemoglobin levels, serum ferritin levels, serum iron levels, TSAT, TIBC, serum albumin levels, CRP and energy consumption (kcal/week) were included in the model as multivariate variables. Backward stepwise logistic regression (ROC) analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable undergoing hemodialysis

Exclusion Criteria:

* Patients those who refused to join present study, and those who could not complete the questionnaires by themselves, and the patients with chronic hepatitis B or C were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study subjects were the patients undergoing HD.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Measurement of depression status | day 1
  Using The Beck Depression Inventory

SECONDARY OUTCOMES:
The values of serum ferritin | day 1
  Measuring serum ferritin levels as iron metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Mizuno-Matsumoto, Ph.D, Study Director — Graduate School of Applied Informatics, University of Hyogo

IPD SHARING:
Plan to Share IPD: No